CLINICAL TRIAL: NCT05935943
Title: Reliability and Validity of the Spinal Cord Injury Secondary Conditions Scale Among the Turkish Population With Spinal Cord Injury
Brief Title: Reliability and Validity of the Spinal Cord Injury Secondary Conditions Scale
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Akpınar, Assoc Prof MD, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: FSMEAH-KAEK 2023/22
Record Dates: First submitted 2023-06-20; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Spinal Cord Injuries; Reliability; Validity
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
People living with spinal cord injury (SCI) experience a range of secondary health conditions that impact their quality of lives. The Spinal Cord Injury Secondary Conditions Scale (SCI-SCS) is a 16-item questionnaire that assess secondary health conditions in persons with SCI. The total score of SCI-SCS range from 0 to 48 and is derived by adding the scores for each item. Higher scores indicate greater problems with secondary conditions. The investigators aimed to determine the reliability and cross-cultural validation of the Turkish translation of the SCI-SCS.

DETAILED DESCRIPTION:
After translation and back translation of the SCI-SCS, 93 patients between the ages of 18 and 78 years with SCI, American Spinal Injury Association impairment scale grades from A to D and at least 6 months after injury were assessed. Participants rated the SCI-SCS 2-3 day apart, and test-retest agreement was investigated. Factor analysis was done and convergent validity was investigated by correlating the SCI-SCS with the Spinal Cord Injury Spasticity Evaluation Tool (SCI-SET), Functional Ambulation Categories (FAC), 36-Item Short Form Health Survey (SF-36), and Spinal Cord Independence Measure III (SCIM-III).

ELIGIBILITY:
Inclusion Criteria:

Patients between the ages of 18 and 80 years with SCI, American Spinal Injury Association impairment scale grades from A to D and at least 6 months after injury. Those who volunteered to participate in the study.

Exclusion Criteria:

* Patients with SCI for less than 6 months
* Patients with impaired cognitive functions,
* Patients with other neurological diseases,
* Patients with malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18 and 80 years with SCI, American Spinal Injury Association impairment scale grades from A to D and at least 6 months after injury who volunteered to participate in the study were recruited from the inpatient and outpatient rehabilitation unit of an education and research hospital.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Reliability of the Spinal Cord Injury Secondary Conditions Scale | 1 year
  Participants rated the Spinal Cord Injury Secondary Conditions Scale (SCI-SCS) 2-3 day apart, and test-retest agreement was investigated for the reliability.

SECONDARY OUTCOMES:
Validity of the Spinal Cord Injury Secondary Conditions Scale | 1year
  Factor analysis was done and convergent validity was investigated by correlating the SCI-SCS with the Spinal Cord Injury Spasticity Evaluation Tool (SCI-SET), Functional Ambulation Categories (FAC), 36-Item Short Form Health Survey (SF-36), and Spinal Cord Independence Measure III (SCIM-III).

CONTACTS AND LOCATIONS:
Overall Officials: FEYZA UNLU OZKAN, Prof, Study Chair — Fatih Sultan Mehmet Training and Research Hospital; ILKNUR AKTAS, Prof, Study Chair — Fatih Sultan Mehmet Training and Research Hospital; ZEYNEP DEMİR, MD, Study Chair — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Fatih Sultan Mehmet Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalpakjian CZ, Scelza WM, Forchheimer MB, Toussaint LL. Preliminary reliability and validity of a Spinal Cord Injury Secondary Conditions Scale. J Spinal Cord Med. 2007;30(2):131-9. doi: 10.1080/10790268.2007.11753924. PMID 17591225
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Wild D, Grove A, Martin M, Eremenco S, McElroy S, Verjee-Lorenz A, Erikson P; ISPOR Task Force for Translation and Cultural Adaptation. Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes (PRO) Measures: report of the ISPOR Task Force for Translation and Cultural Adaptation. Value Health. 2005 Mar-Apr;8(2):94-104. doi: 10.1111/j.1524-4733.2005.04054.x. PMID 15804318